CLINICAL TRIAL: NCT06253871
Title: A Phase 1/1b Study of IAM1363 in Patients With Advanced Cancers Harboring HER2 Alterations
Brief Title: A Phase 1/1b Study of IAM1363 in HER2 Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Iambic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAM1363-01
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: HER2 Mutation-Related Tumors; HER2; HER2-positive Breast Cancer; HER2 + Breast Cancer; Brain Metastases From Solid Tumors; Brain Metastases From HER2 and Breast Cancer; CNS Metastases; HER2-Positive Solid Tumors; NSCLC (Non-small Cell Lung Cancer); HER2-positive Bladder Cancer; HER2-positive Colorectal Cancer; HER2 + Gastric Cancer; HER2-positive Gastroesophageal Cancer
Keywords: ERBB2 protein, human; Molecular Targeted Therapy; Genes, erbB-2; Receptor, ErbB-2 / antagonists & inhibitors; Neoplasms / drug therapy; HER2 positive; HER2 overexpressing; HER2 altered; Human epidermal growth factor receptor; ErbB Receptors; HER2; brain metastases
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Neoplasms; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose-escalation and dose optimization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IAM1363 Monotherapy (Experimental): Treatment with IAM1363 capsules, dosed orally either once or twice daily in 21-day cycles.
  Interventions: Drug: IAM1363

INTERVENTIONS:
Drug: IAM1363 — Oral, immediate release capsules of IAM1363

SUMMARY:
This is a Phase 1/1b open-label, multi-center dose escalation and dose optimization study designed to evaluate the safety and preliminary efficacy of IAM1363 in participants with advanced cancers that harbor HER2 alterations.

DETAILED DESCRIPTION:
This is a Phase 1/1b open-label, multi-center study, designed to evaluate IAM1363 in participants with advanced cancers that harbor HER2 alterations.

This study consists of the following 3 parts, which are described in further detail below:

* Part 1 (Monotherapy Dose Escalation)
* Part 2 (Dose Optimization)
* Part 3 (Simon 2-Stage Evaluation)

Part 1 will enroll participants with a confirmed, relapsed/refractory malignancy with documented diagnosis of HER2 alterations including participants with brain metastases. Once a provisional maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) has been determined, Part 2 will enroll additional cohorts to optimize dose selection and to further evaluate the safety and preliminary efficacy of IAM1363. Following completion of Dose Optimization, Part 3 will be opened to enroll tumor-specific cohorts utilizing a Simon 2-Stage Minimax Design to evaluate IAM1363 at the selected dose(s).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Have relapsed/refractory HER2-altered malignancy
* Have progression of disease after the last systemic therapy, or be intolerant of last systemic therapy
* Have radiographically measurable disease by RECIST v1.1 and/or RANO-BM
* Eastern Cooperative Oncology Group (ECOG) performance score 0-1
* Have adequate baseline hematologic, liver and renal function
* Have left ventricular ejection fraction (LVEF) ≥ 50%

Key Exclusion Criteria:

* Clinically significant cardiac disease
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2. Exception: Patients with well-controlled HIV (e.g., CD4 >350/mm3 and undetectable viral load) are eligible
* Current active liver disease including hepatitis A, hepatitis B , or hepatitis C
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate absorption
* Uncontrolled diabetes
* History of solid organ transplantation
* History of Grade ≥2 CNS hemorrhage, or any CNS hemorrhage within 28 days before C1D1
* Patients requiring immediate local therapy for brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) (Part 1 only) | 21 days
  Incidence and severity of DLTs during the first cycle of treatment in participants in Part 1
Incidence and severity of adverse events (AEs) (Parts 1 and 2 only) | Through 30 days after the last dose of study drug
  Incidence of treatment emergent AEs (TEAEs) and serious adverse events (SAEs) in participants in Parts 1 and 2
Pharmacokinetic (PK) parameters (Parts 1 and 2 only) | Up to 42 days
  PK parameters in participants in Parts 1 and 2. Includes but is not limited to assessment of maximum concentration (Cmax).
Pharmacokinetic (PK) parameters (Parts 1 and 2 only) | Up to 42 days
  PK parameters in participants in Parts 1 and 2. Includes but is not limited to assessment of time to maximum concentration (Tmax).
Pharmacokinetic (PK) parameters (Parts 1 and 2 only) | Up to 42 days
  PK parameters in participants in Parts 1 and 2. Includes but is not limited to assessment of area under the curve (AUC).
Confirmed objective response rate (cORR) (Part 3 only) | Through study completion, estimated as 46 months
  Percentage of participants in Part 3 who achieve a confirmed objective response (complete response [CR] + partial response [PR]) per the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
Confirmed central nervous system ORR (CNS-cORR) (Part 3 Only) | Through study completion, estimated as 46 months
  Percentage of participants in Part 3 who achieve a confirmed CNS-cORR (CNS-CR + CNS-PR) per the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) Criteria

SECONDARY OUTCOMES:
Incidence and severity of clinical laboratory abnormalities | Through 30 days after the last dose of study drug
  Incidence and severity of clinical laboratory abnormalities
Incidence of electrocardiogram (ECG) abnormalities | Through 30 days after the last dose of study drug
  Incidence of ECG abnormalities, as measured using standard ECG parameters, including respiratory rate, pulse rate, QT intervals, and QRS duration.
cORR (Parts 1 and 2 only) | Through study completion, estimated as 46 months
  Percentage of participants in Parts 1 and 2 with cORR (CR + PR) per RECIST v1.1
Best overall response (BoR) rate | Through study completion, estimated as 46 months
  BoR defined as the best response per RECIST v1.1 across all assessments
Duration of response (DoR) | Through study completion, estimated as 46 months
  DoR defined as the time between the first confirmed objective response per RECIST v1.1 and date of disease progression per RECIST v1.1 or death due to any cause
Disease control rate (DCR) | Through study completion, estimated as 46 months
  DCR defined as the percentage of participants who achieve CR or PR, or stable disease (SD) per RECIST v1.1 consecutively for 3 months
Clinical benefit rate (CBR) | Through study completion, estimated as 46 months
  CBR defined as the percentage of participants who achieve CR, PR, or SD per RECIST v1.1
Progression-free survival (PFS) | Through study completion, estimated as 46 months
  PFS defined as the number of months from the date of first study treatment administration to the earliest of documented progressive disease per RECIST v1.1 or death without prior progression
Overall survival (OS) | Through study completion, estimated as 46 months
  OS defined as the number of months from the date of first study treatment administration to the date of death, irrespective of cause
Incidence and severity of AEs (Part 3 Only) | Through 30 days after the last dose of study drug
  Incidence and severity of treatment emergent AEs and SAEs in participants in Part 3
PK parameters (Part 3 only) | Up to 42 days
  PK parameters in participants in Part 3. Includes but is not limited to assessment of maximum concentration (Cmax).
PK parameters (Part 3 only) | Up to 42 days
  PK parameters in participants in Part 3. Includes but is not limited to assessment of time to maximum concentration (Tmax).
PK parameters (Part 3 only) | Up to 42 days
  PK parameters in participants in Part 3. Includes but is not limited to assessment of area under the curve (AUC).
Anti-tumor activity against CNS/brain metastases | Through study completion, estimated as 46 months
  Anti-tumor response based on RANO-BM Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Iambic Therapeutics, Inc., Senior Medical Director, Study Director — Iambic Therapeutics, Inc
Locations (45):
- United States (28):
  - UCSD Moores Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - START - Midwest Cancer Research Center, Grand Rapids, Michigan
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - RUTGERS Cancer Institute, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute, Portland, Oregon
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - NEXT Oncology - Austin, Austin, Texas
  - NEXT Oncology - Dallas, Dallas, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center - University of Texas, Houston, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Oncology - Virginia Cancer Specialists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- France (3):
  - Centre Georges François Leclerc, Dijon
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse (IUCT) Oncopole Institut Claudius Regaud ", Toulouse
- Ireland (3):
  - The START center Dublin, Dublin, Dublin
  - Cork University Hospital, Wilton, Cork
  - St. Vincent's University Hospital, Dublin
- Azienda Ospedaliero Universitaria Careggi - Largo Giovanni Alessandro Brambilla 3, Florence, Italy
- Netherlands Cancer Institute-Antoni van Leeuwenhoek, Amsterdam, Netherlands
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitario Vall dHebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid CIOCC, Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia (INCLIVA), Valencia